CLINICAL TRIAL: NCT00731549
Title: A 52-week, Multicenter, Open-label Study to Evaluate the Effectiveness of Aripiprazole Intramuscular Depot as Maintenance Treatment in Patients With Schizophrenia
Brief Title: Intramuscular Depot Formulation of Aripiprazole as Maintenance Treatment in Patients With Schizophrenia
Acronym: ASPIRE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 31-08-248
Record Dates: First submitted 2008-08-05; First posted 2008-08-11 (Estimated); Results first posted 2014-11-11 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Schizophrenia
Keywords: Aripiprazole; IM Depot; Schizophrenia; Intramuscular
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Active Treatment of aripiprazole IM depot (300mg or 400mg)
  Interventions: Drug: Aripiprazole IM Depot

INTERVENTIONS:
Drug: Aripiprazole IM Depot — 300mg or 400mg
  Other Names: Oral Aripiprazole

SUMMARY:
To evaluate the overall effectiveness of aripiprazole intramuscular (IM) depot as maintenance treatment in patients with schizophrenia.

DETAILED DESCRIPTION:
This will be an open-label, uncontrolled study which will enroll subjects from Phase 4 of Study 31-07-246 and Phase 3 of Study 31- 07-247 and new subjects not participating in Studies 246/247. The treatment history of subjects prior to enrollment in the open-label study will vary according to the design of the pivotal double-blind study (i.e., 31-07-246 or 31-07-247).

This open-label study will be comprised of phases similar to the pivotal double-blind studies (i.e., Studies 246/247): a screening phase (if applicable), a conversion phase (Phase 1, if applicable), an oral stabilization phase (Phase 2), and an IM depot open-label maintenance phase (Phase 3). Phase 3 will be a 52-week treatment period with a 26-week follow-up period.

During Phase 3 (the open-label maintenance phase) oral aripiprazole rescue medication will be allowed for subjects who do not meet stability criteria or meet the criteria for impending relapse/exacerbation of psychotic symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are able to provide written informed consent and/or consent obtained from a legally acceptable representative (as require by IRB/IEC), prior to the initiation of any protocol-required procedures.
* Male and female subjects 18 to 65 years of age, inclusive, at time of informed consent.
* Subjects who complete Studies 246/247 or who withdrew from the double-blind maintenance phase of either study (Phase 4 of Study 246 or Phase 3 of Study 247), or new subjects not participating in Studies 246/247.
* # Subjects who, in the investigator's judgment, require chronic treatment with an antipsychotic medication.
* Subjects able to understand the nature of the study and follow protocol requirements, including the prescribed dosage regimens, tablet ingestion, IM depot injection, discontinuation of prohibited concomitant medications, who can read and understand the written word in order to complete patient-reported outcomes measures, and who can be reliably rated on assessment scales.

Exclusion Criteria:

* Subjects with a current DSM-IV-TR diagnosis other than schizophrenia, including schizoaffective disorder, major depressive disorder, bipolar disorder, delirium, dementia, amnestic or other cognitive disorders. Also, subjects with borderline, paranoid, histrionic, schizotypal, schizoid or antisocial personality disorder.
* Subjects with schizophrenia that are considered resistant/refractory to antipsychotic treatment by history or response only to clozapine.
* Subjects with a significant risk of violent behavior or a significant risk of committing suicide based on history or investigator's judgment.
* Subjects who currently meet DSM-IV-TR criteria for substance dependence; including alcohol and benzodiazepines, but excluding caffeine and nicotine, or two positive drug screens for cocaine.
* Subjects who are known to be allergic, intolerant, or unresponsive to prior treatment with aripiprazole or other quinolinones.
* Subjects with a history of hypersensitivity to antipsychotic agents.
* Subjects with a history of neuroleptic malignant syndrome or clinically significant tardive dyskinesia at screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1081 (Actual)
Dates: Start 2008-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (179):
- United States (82):
  - Chandler, Arizona
  - Anaheim, California
  - Cerritos, California
  - Chino, California
  - Escondido, California
  - Garden Grove, California
  - Glendale, California
  - Imperial, California
  - La Habra, California
  - Los Angeles, California
  - National City, California
  - Oceanside, California
  - Orange, California
  - Pasadena, California
  - Pico Rivera, California
  - San Bernardino, California
  - San Diego, California
  - Study Site, San Diego, California
  - Sherman Oaks, California
  - Torrance, California
  - Highlands Ranch, Colorado
  - Norwalk, Connecticut
  - Washington D.C., District of Columbia
  - Bradenton, Florida
  - Coral Springs, Florida
  - Doral, Florida
  - Gainesville, Florida
  - Hollywood, Florida
  - Kissimmee, Florida
  - Maitland, Florida
  - Miami, Florida
  - Orange City, Florida
  - Orlando, Florida
  - Plantation, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Hoffman Estates, Illinois
  - Oak Brook, Illinois
  - Indianapolis, Indiana
  - Baton Rouge, Louisiana
  - Lake Charles, Louisiana
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Columbia, Maryland
  - Flowood, Mississippi
  - Kansas City, Missouri
  - St Louis, Missouri
  - North Platte, Nebraska
  - Albuquerque, New Mexico
  - Buffalo, New York
  - Cedarhurst, New York
  - Holliswood, New York
  - Jamaica, New York
  - New York, New York
  - Rochester, New York
  - Hickory, North Carolina
  - Winston-Salem, North Carolina
  - Canton, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Garfield Heights, Ohio
  - Middleburg Heights, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Allentown, Pennsylvania
  - Jenkintown, Pennsylvania
  - Media, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Sellersville, Pennsylvania
  - Charleston, South Carolina
  - Johnson City, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - DeSoto, Texas
  - Richmond, Virginia
  - Bellevue, Washington
  - Bothell, Washington
  - Spokane, Washington
  - Milwaukee, Wisconsin
- Argentina (4):
  - Buenos Aires
  - Cordoba, Cordoba
  - La Plata, Buenos Aires
  - Mendoza
- Australia (6):
  - Dandenong, Victoria
  - Epping, Victoria
  - Frankston, Victoria
  - Fremantle, Western Australia
  - Glenside, SA
  - Melbourne
- Innsbruck, Austria
- Bruges, Belgium
- Bulgaria (10):
  - Burgas
  - Lovech
  - Pazardzhik
  - Pleven
  - Plovdiv
  - Radnevo
  - Rousse
  - Sofia
  - Varna
  - Veliko Tarnovo
- Chile (2):
  - San Bernardo, Santiago
  - Santiago
- Zagreb, Croatia
- Estonia (3):
  - Jämejala
  - Tallinn
  - Tartu
- Helsinki, Finland
- France (3):
  - Élancourt
  - Rennes
  - Saint-Nazaire
- Hungary (4):
  - Baja
  - Balassagyarmat
  - Cegléd
  - Győr
- India (7):
  - Ahmedabad, Gujarat
  - Bangalore, Karnataka
  - Chennai, Tamil Nadu
  - Kanpur
  - Mangalore
  - Pune
  - Tirupati
- Malaysia (3):
  - Kuala Lumpur, Kuala Lumpur
  - Tanjong Rambutan, Perak
  - Kuala Selangor
- Mexico (5):
  - Guadalajara, Jalisco
  - Mexico City, Mexico City
  - Monterrey, Nuevo León
  - San Luis Potosí City, San Luis Potosí
  - Culiacán, Sinaloa
- Norway (2):
  - Ålesund
  - Klepp stasjon
- Philippines (4):
  - Bataan, Central Luzon
  - Mandaluyong, NCR
  - Quezon City, NCR
  - Iloilo City, Western Visayas
- Poland (9):
  - Bełchatów
  - Bialystok
  - Bydgoszcz
  - Choroszcz
  - Krakow
  - Leszno
  - Pruszków
  - Sosnowiec
  - Wroclaw
- San Juan, Puerto Rico
- Romania (6):
  - Arad
  - Bucharest
  - Cluj-Napoca
  - Craiova
  - Oradea
  - Piteşti
- Russia (5):
  - Lipetsk
  - Moscow
  - Nizhny Novgorod
  - Saint Petersburg
  - Smolensk
- Serbia (2):
  - Belgrade
  - Kragujevac
- Slovakia (5):
  - Košice
  - Liptovský Mikuláš
  - Prešov
  - Rimavská Sobota
  - Svidník
- South Africa (2):
  - Pretoria, Gauteng
  - Cape Town, Western Province
- South Korea (5):
  - Busan
  - Deajeon
  - Gwangju
  - Joong-gu, Incheon
  - Seoul
- Barcelona, Spain
- Taiwan (2):
  - Tainan
  - Taipei
- Thailand (2):
  - Muang, Chiangmai
  - Bangkok

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This open label Phase 3 study enrolled participants from the maintenance phase of study NCT00705783 (31-07-246) and study NCT00706654 (31-07-247) and new participants. Participants received aripiprazole intramuscular (IM) depot as maintenance treatment.
Pre-assignment Details: Study comprised of screening phase (applicable if enrolled late/new participants/received antipsychotic treatment other than aripiprazole), conversion phase (Phase 1, to convert from other antipsychotics to aripiprazole), oral stabilization phase (Phase 2-aripiprazole 10-30 mg), and open-label IM phase (Phase 3-aripiprazole 400 mg IM depot).
Groups:
- Aripiprazole 400/300 mg IM Depot: Participants received open-label aripiprazole 400/300 mg IM depot into gluteal muscle every 4 weeks for a maximum of 52 weeks. Flexible dosing with apipiprazole 300 mg and 400 mg is permitted in order to maximize retention of participants. Partipants also received supplemental oral aripiprazole (10 mg to 20 mg daily) for the first two weeks to maintain therapeutic plasma concentrations.
Period: Overall Study
Arm/Group | Aripiprazole 400/300 mg IM Depot
Started | 1081
Completed | 858
Not Completed | 223
Not completed — Lost to Follow-up | 19
Not completed — Met withdrawal criteria | 24
Not completed — Physician Decision | 16
Not completed — Withdrawal by Subject | 89
Not completed — Protocol deviation | 1
Not completed — Adverse Event | 31
Not completed — Lack of efficacy with AE | 37
Not completed — Lack of efficacy without AE | 6

BASELINE CHARACTERISTICS:
Arm/Group | Aripiprazole 400/300 mg IM Depot
Number analyzed (Participants) | 1081
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.2 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 439
  Male | 642

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Stable Participants at Baseline Who Remained Stable at Endpoint (Last Visit).
Description: "Stable" was defined as meeting all of the following criteria: Outpatient status; Positive and negative syndrome scale (PANSS) total score ≤ 80; Lack of specific psychotic symptoms on the PANSS as measured by a score of ≤ 4 on each of the following items (possible scores of 1 to 7 for each item): 1) conceptual disorganization 2) suspiciousness 3) hallucinatory behavior 4) unusual thought content; Clinical Global Impression of Severity (CGI-S) ≤ 4 (moderately ill); and Clinical Global Impression for Severity of Suicidality (CGI-SS) ≤ 2 (mildly suicidal) on Part 1 and ≤ 5 (minimally worsened) on Part 2. The percentage of stable participants at baseline who remain stable at endpoint (last visit) is described here.
Time Frame: Baseline to Week 52/Last visit
Population: All participants who entered Phase 3 and have at least one post-baseline efficacy evaluation in Phase 3 are included. N defines number of stable participants at baseline who were evaluated at the specified trial week.
Measure: Number; unit: Percentage of participants
Arm/Group | Aripiprazole 400/300 mg IM Depot
Number analyzed (Participants) | 1081
Percentage of participants
  Baseline (N=1075) | 100
  Week 2 (N=1023) | 99.02
  Week 4 (N=1045) | 99.14
  Week 8 (N=1009) | 98.51
  Week 12 (N=988) | 97.47
  Week 16 (N=951) | 98.42
  Week 20 (N=919) | 98.15
  Week 24 (N=880) | 99.20
  Week 28 (N=854) | 98.95
  Week 32 (N=838) | 99.16
  Week 36 (N=814) | 99.26
  Week 40 (N=807) | 99.50
  Week 44 (N=784) | 99.11
  Week 48 (N=751) | 99.20
  Week 52 (N=671) | 98.96
  Last visit (N=1072) | 94.96

2. Secondary Outcome: Percentage of Participants Meeting Exacerbation of Psychotic Symptoms/Impending Relapse Criteria.
Description: "Impending relapse criteria" was defined as meeting all the following criteria: 1) Clinical Global Impression of Improvement (CGI-I) ≥ 5 (minimally worse), AND an increase to score of >4 and absolute increase of ≥ 2 on the individual PANSS items (conceptual disorganization, hallucinatory behavior, suspiciousness, unusual thought content); or an increase to score >4 and absolute increase of ≥ 4 on the combined 4 PANSS items on any of these PANSS items (conceptual disorganization, hallucinatory behavior, suspiciousness, unusual thought content) OR 2) Hospitalization due to worsening of psychotic symptoms, but excluding hospitalization for psychosocial reasons, OR 3) CGI-SS score of 4 (severely suicidal) or 5 (attempted suicide) on Part 1 and/or 6 (much worse) or 7 (very much worse) on Part 2, OR 4) Violent behavior resulting in clinically relevant self-injury, injury to another person, or property damage.
Time Frame: Weeks 2,4,8,12,16,20,24,28,32,36,40,44,48,52, and Last visit (upto 4 weeks ± 3 days after completion or withdrawal)
Population: All participants who entered Phase 3 and have at least one post-baseline efficacy evaluation in Phase 3 are included. N defines number of participants evaluated at the specified trial week.
Measure: Number; unit: Percentage of participants
Arm/Group | Aripiprazole 400/300 mg IM Depot
Number analyzed (Participants) | 1081
Percentage of participants
  Week 2 (N=1028) | 0.49
  Week 4 (N=1049) | 0.48
  Week 8 (N=1011) | 0.79
  Week 12 (N=988) | 1.52
  Week 16 (N=948) | 0.84
  Week 20 (N=920) | 1.09
  Week 24 (N=883) | 0.45
  Week 28 (N=857) | 0.58
  Week 32 (N=838) | 0.36
  Week 36 (N=814) | 0.25
  Week 40 (N=808) | 0.25
  Week 44 (N=783) | 0.26
  Week 48 (N=750) | 0.27
  Week 52 (N=668) | 0.30
  Last visit (N=1079) | 4.17
  Overall (N=1079) | 8.25

3. Secondary Outcome: Percentage of Participants Achieving Remission.
Description: Remission is defined as a score of ≤ 3 on each of the following specific PANSS items, maintained for a period of six months: delusions, unusual thought content, hallucinatory behavior, conceptual disorganization, mannerisms/posturing, blunted affect, social withdrawal, and lack of spontaneity.
Time Frame: Overall remission from Weeks 2,4,8,12,16,20,24,28,32,36,40,44,48 and 52
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Aripiprazole 400/300 mg IM Depot
Number analyzed (Participants) | 1081
Percentage of participants | 51.7

4. Secondary Outcome: Percentage of Participants Stable at Baseline and Remaining Stable at Week 28.
Description: "Stable" was defined as meeting all of the following criteria: Outpatient status; PANSS total score ≤ 80; Lack of specific psychotic symptoms on the PANSS as measured by a score of ≤ 4 on each of the following items (possible scores of 1 to 7 for each item): 1) conceptual disorganization 2) suspiciousness 3) hallucinatory behavior 4) unusual thought content; Clinical Global Impression of Severity (CGI-S) ≤ 4 (moderately ill); and Clinical Global Impression for Severity of Suicidality (CGI-SS) ≤ 2 (mildly suicidal) on Part 1 and ≤ 5 (minimally worsened) on Part 2. The percentage of stable participants at baseline who remain stable at Week 28 is described here.
Time Frame: Baseline to Week 28
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Aripiprazole 400/300 mg IM Depot
Number analyzed (Participants) | 1081
Percentage of participants
  Baseline (N=1075) | 100
  Week 28 (N=854) | 98.95

5. Secondary Outcome: Percentage of Participants With Time to First Exacerbation of Psychotic Symptoms/Impending Relapse.
Description: Participants who first time meet relapse criteria were considered as having an event at date of exacerbation of psychotic symptoms/impending relapse. Time to first event was calculated as the earliest date of meeting one of relapse criteria. Limited concurrent treatment with oral aripiprazole was permitted as rescue therapy.
Time Frame: Baseline to Week 52
Population: All participants who entered Phase 3 and have at least one post-baseline efficacy evaluation in Phase 3 are included. Number of participants analyzed had available assessments for evaluation of exacerbation of psychotic symptoms/impending relapse.
Measure: Number; unit: Percentage of participants
Arm/Group | Aripiprazole 400/300 mg IM Depot
Number analyzed (Participants) | 1079
Percentage of participants | 8.2

6. Secondary Outcome: Mean Change From Baseline to Endpoint (Last Visit) in Positive and Negative Syndrome Scale (PANSS) Total Score.
Description: PANSS total score (range 30-210) is the sum of the rating scores for 7 positive scale items, 7 negative scale items and 16 general psychopathology scale items from the PANSS scale. PANSS positive subscale score (range 7-49) is the sum of the rating scores for the 7 positive scale items from the PANSS scale. PANSS negative subscale score (range 7-49) is the sum of the rating scores for the 7 negative scale items from the PANSS scale. The severity of each scale is rated on a 7-point scale, with a score of 1 indicating the absence of symptoms and a score of 7 indicating extremely severe symptoms.
Time Frame: Baseline, Weeks 12, 24, 52 and last visit
Population: All participants who entered Phase 3 and have at least one post-baseline efficacy evaluation in Phase 3 are included. Number of participants analyzed with baseline or at least one postbaseline assessment are included here.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole 400/300 mg IM Depot
Number analyzed (Participants) | 1081
Units on a scale
  Week 12 (N=987) | -1.69 (6.21)
  Week 24 (N=882) | -2.55 (7.08)
  Week 52 (N=669) | -3.55 (7.75)
  Last visit (N=1078) | -1.72 (10.21)

7. Secondary Outcome: Mean Change From Baseline in Clinical Global Impression of Severity (CGI-S) Score.
Description: To assess CGI-S, the rater or physician will answer the following question: "Considering your total clinical experience with this particular population, how mentally ill is the participant at this time?" Response choices include: 0 = not assessed; 1 = normal, not ill at all; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill participants.
Time Frame: Baseline, Weeks 12, 24, 52 and last visit
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole 400/300 mg IM Depot
Number analyzed (Participants) | 1081
Units on a scale
  Week 12 (N=987) | -0.11 (0.52)
  Week 24 (N=883) | -0.17 (0.53)
  Week 52 (N=668) | -0.24 (0.56)
  Last visit (N=1079) | -0.14 (0.70)

8. Secondary Outcome: Mean Change From Baseline to Endpoint in PANSS Positive and Negative Subscales.
Description: PANSS positive subscale score (range 7-49) is the sum of the rating scores for the 7 positive scale items from the PANSS scale. Positive subscale consists of 7 positive symptom constructs: delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, and hostility). PANSS negative subscale score (range 7-49) is the sum of the rating scores for the 7 negative scale items from the PANSS scale. Negative subscale consists of 7 negative symptom constructs: blunted affect, emotional withdrawal, poor rapport, passive pathetic withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation, stereotyped thinking). The severity of each scale is rated on a 7-point scale, with a score of 1 indicating the absence of symptoms and a score of 7 indicating extremely severe symptoms.
Time Frame: Baseline, Weeks 12, 24, 52 and last visit
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole 400/300 mg IM Depot
Number analyzed (Participants) | 1081
Units on a scale
  Week 12 positive subscale score (N=987) | -0.42 (2.11)
  Week 24 positive subscale score (N=882) | -0.68 (2.26)
  Week 52 positive subscale score (N=669) | -1.04 (2.53)
  Last visit positive subscale score (N=1078) | -0.49 (3.38)
  Week 12 negative subscale score (N=987) | -0.40 (2.40)
  Week 24 negative subscale score (N=882) | -0.53 (2.52)
  Week 52 negative subscale score (N=669) | -0.80 (2.94)
  Last visit negative subscale score (N=1078) | -0.46 (3.19)

9. Secondary Outcome: Mean Clinical Global Impression of Improvement (CGI-I) Score.
Description: To assess CGI-I the rater or physician will rate the participant's total improvement whether or not it is due entirely to drug treatment. All responses will be compared to the participants condition at baseline. Response choices include: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse.
Time Frame: Weeks 2, 4, 12, 24, 52 and last visit
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole 400/300 mg IM Depot
Number analyzed (Participants) | 1081
Units on a scale
  Baseline (N=1081) | 3.48 (0.82)
  Week 2 (N=1026) | 3.52 (0.85)
  Week 4 (N=1049) | 3.49 (0.86)
  Week 12 (N=987) | 3.42 (0.92)
  Week 24 (N=882) | 3.33 (0.98)
  Week 52 (N=669) | 3.25 (0.99)
  Last visit (N=1079) | 3.35 (1.10)

10. Secondary Outcome: Percentage of Participants Who Discontinued Due to All Causes.
Description: Participants who discontinued due to any cause were noted. Limited concurrent treatment with oral aripiprazole was permitted as rescue therapy.
Time Frame: Baseline to Week 52
Population: All participants who entered Phase 3 and have at least one post-baseline efficacy evaluation in Phase 3 are included.
Measure: Number; unit: Percentage of participants
Arm/Group | Aripiprazole 400/300 mg IM Depot
Number analyzed (Participants) | 1081
Percentage of participants | 20.6

ADVERSE EVENTS:
Time Frame: Phase 3 Week 1 to Week 52/Early termination.
Description: All participants who had received at least one dose of aripiprazole IM depot were included in safety analysis.
Arm/Group | Aripiprazole 400/300 mg IM Depot
Serious Adverse Events (participants affected / at risk) | 95/1081
Other Adverse Events (participants affected / at risk) | 254/1081
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole 400/300 mg IM Depot (N=1081)
Anaemia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiac failure acute (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 2
Open angle glaucoma (Eye disorders) | 1
Uveitis (Eye disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Stomach mass (Gastrointestinal disorders) | 1
Facial pain (General disorders) | 1
Sudden death (General disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 2
Bronchitis (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 2
Gangrene (Infections and infestations) | 1
Genital candidiasis (Infections and infestations) | 1
Hepatitis viral (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Pilonidal cyst (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 4
Respiratory tract infection (Infections and infestations) | 1
Syphilis (Infections and infestations) | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Intentional overdose (Injury, poisoning and procedural complications) | 2
Multiple injuries (Injury, poisoning and procedural complications) | 1
Liver function test abnormal (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tongue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Convulsion (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Ruptured cerebral aneurysm (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Adjustment disorder (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
Hallucination, auditory (Psychiatric disorders) | 2
Homicidal ideation (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 15
Schizoaffective disorder (Psychiatric disorders) | 1
Schizophrenia (Psychiatric disorders) | 21
Schizophrenia, paranoid type (Psychiatric disorders) | 5
Suicidal ideation (Psychiatric disorders) | 2
Suicide attempt (Psychiatric disorders) | 3
Menorrhagia (Reproductive system and breast disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Arteriosclerosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole 400/300 mg IM Depot (N=1081)
Nasopharyngitis (Infections and infestations) | 76
Headache (Nervous system disorders) | 82
Anxiety (Psychiatric disorders) | 73
Insomnia (Psychiatric disorders) | 71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No